CLINICAL TRIAL: NCT01986569
Title: A Phase III, Open Label, Non-randomized, Single Center Study to Evaluate Diagnostic Accuracy and Safety of Fluorine-18 (18F) Fluoroestradiol PET/CT in the Assessment of ER Status of Recurrent or Metastatic Lesions in Patients With Breast Cancer
Brief Title: Diagnostic Accuracy and Safety Study of FES PET/CT in Assessment of ER Status of Recurrent or Metastatic Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Dae Hyuk Moon, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FES13001
Record Dates: First submitted 2013-11-12; First posted 2013-11-18 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Recurrent Breast Cancer; Stage IV Breast Cancer
Keywords: Fluoroestradiol (FES); PET/CT scan; Estrogen Receptor; Recurrent breast cancer; Stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- [18F]fluoroestradiol (FES) (Experimental): The injectable radioactive dose of 111-222 megabecquerel. One single IV injection over 1-2 min. [18F]FES PET/CT for imaging.
  Interventions: Drug: [18F]fluoroestradiol (FES)

INTERVENTIONS:
Drug: [18F]fluoroestradiol (FES) — [18F]FES PET/CT will be performed 90 min (± 10 min) after administration of [18F]FES. Patients will undergo core needle biopsy or surgery within 15 days after [18F]FES PET; or patients will undergo core needle biopsy within 30 days before [18F]FES PET. Experienced pathologists will determine metastatic/recurrent disease, and tumor histology including IHC. Patient will undergo surgery, radiation therapy or systemic therapy according to the results of staging workup, histology and biomarkers.

SUMMARY:
The standard diagnostic workup for recurrent or metastatic breast cancer includes biopsy and determination of tumor estrogen status according to National Comprehensive Cancer Network and European Society for Medical Oncology. Immunohistochemistry (IHC) is currently the most commonly used method for determining ER status. A investigational imaging tracer named 16-alpha-[18F]-fluoro-17-beta-estradiol, or [18F]fluoroestradiol ([18F]FES) acts similarly in vivo to estradiol and binds to estrogen receptors (ERs). Previous studies in human have shown the efficacy of [18F]FES PET in detecting ER positive breast cancer without any observed toxicity. The investigators hypothesized that [18F]FES PET imaging can noninvasively assess ER status in recurrent or metastatic breast cancer lesion . In this study, a positive and negative percent agreement between IHC and [18F]FES will be determined.

ELIGIBILITY:
Inclusion Criteria:

* A patient will be enrolled if the patient meets the following inclusion criteria

  1. Patient is ≥19 years of age and male or female of any race/ethnicity
  2. Patients has first recurrence or stage IV disease by American Joint Committee on Cancer tumor-node-metastasis staging system for breast cancer
  3. Patients had histologically confirmed invasive primary breast carcinoma and the documented results of histology are available.
  4. Patients are scheduled to undergo core needle biopsy or surgery for histological confirmation and determination of ER status of recurrent or distant metastatic cancer within 15 days after [18F]FES PET; or patients already underwent core needle biopsy of recurrent or distant metastatic cancer within 30 days before [18F]FES PET and biopsy specimens are available for determination of ER status.
  5. Discontinuation of selective ER blocking agents including tamoxifen or fulvestrant for at least 60 days prior to [18F]FES PET
  6. Eastern Cooperative Oncology Group (ECOG) performance status of ≤2

Exclusion Criteria:

* A patient will be excluded from this study if the patient does not full fulfill the inclusion criteria, or if any of the following conditions are observed

  1. Patient or patient's legally acceptable representative do not provide written informed consent
  2. The recurrent or metastatic lesion scheduled to undergo biopsy is located in breast, liver, ovary, uterus, or bone
  3. Female patient is pregnant or nursing. Exclusion of the possibility of pregnancy is made by one of the following: 1) woman is physiologically post menopausal (cessation of menses for more than 2 years), 2) woman is surgically sterile (has had a documented bilateral oophorectomy and/or documented hysterectomy, or 3) if the woman is of childbearing potential, a urine pregnancy test performed within 24 hours immediately prior to administration of [18F]FES has to be negative and the women is advised to apply contraceptive measures during her participation in this study
  4. Adjuvant chemotherapy within 3 weeks prior to [18F]FES PET.
  5. Radiation therapy or immuno/biologic therapy is scheduled to be given to patient before the histologic confirmation by biopsy or [18F]FES PET.
  6. Concurrent severe and/or uncontrolled and/or unstable medical disease other than cancer (e.g. congestive heart failure, acute myocardial infarction, severe pulmonary disease, chronic renal or hepatic disease which could compromise participation in the study) in the judgment of the investigator.
  7. Patient is a relative of the investigator, student of the investigator or otherwise dependent
  8. Patient has any other condition or personal circumstances that, in the judgment of the investigator, might interfere with the collection of complete data
  9. Patient has been involved in an investigative, radioactive research procedure within 7 days prior to registration

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2013-11; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
lesion-level positive and negative percent agreement between qualitative [18F]FES PET interpretation and reference IHC testing | up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Dae Hyuk Moon, MD. PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Chae SY, Ahn SH, Kim SB, Han S, Lee SH, Oh SJ, Lee SJ, Kim HJ, Ko BS, Lee JW, Son BH, Kim J, Ahn JH, Jung KH, Kim JE, Kim SY, Choi WJ, Shin HJ, Gong G, Lee HS, Lee JB, Moon DH. Diagnostic accuracy and safety of 16alpha-[18F]fluoro-17beta-oestradiol PET-CT for the assessment of oestrogen receptor status in recurrent or metastatic lesions in patients with breast cancer: a prospective cohort study. Lancet Oncol. 2019 Apr;20(4):546-555. doi: 10.1016/S1470-2045(18)30936-7. Epub 2019 Mar 4. PMID 30846327
- See also: Genetics Home Reference related topics; breast cancer — http://ghr.nlm.nih.gov/condition/breast-cancer
- See also: MedlinePlus related topics; Breast cancer — http://www.nlm.nih.gov/medlineplus/breastcancer.html